CLINICAL TRIAL: NCT06174883
Title: Folic Acid-fortified Iodized Salt and Serum Folate Concentration in Reproductive-aged Women of Rural India
Brief Title: Salt-FA to Increase Folate Levels
Status: Completed | Type: Observational
Sponsor: Hydrocephalus and Neuroscience Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DFS-1-2022
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Neural Tube Defects; Folic Acid Deficiency; Spina Bifida; Anencephaly-Spina Bifida
MeSH Terms: conditions — Neural Tube Defects; Folic Acid Deficiency; Spinal Dysraphism; Neural tube defects X-linked

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Folic acid fortified iodized salt — addition of folic acid to iodized salt to be consumed daily and assess rise in serum folate levels.

SUMMARY:
Question: How effective is folic acid-fortified iodized salt in increasing serum folate concentrations among non-pregnant and non-lactating women of reproductive age? Hypothesis: Folic acid-fortified iodized salt can increase serum folate levels and serve as a policy consideration in salt fortification with both iodine and folic acid to reduce serious and fatal birth defects.

DETAILED DESCRIPTION:
Salt is an ideal vehicle for fortification because its universal consumption and often centrally processed with established distribution channels. Over 70% of households globally have access to iodized salt. Considering the success of salt iodization, it is logical to use the existing infrastructure to provide folic acid through this dietary mechanism.

AIM:To assess increase in blood folate concentrations among women of reproductive age after they consume folic acid-fortified iodized salt.

OBJECTIVES :

1. To examine the effect of consumption of salt fortified with folic acid on serum/plasma folate concentrations among women of reproductive age.
2. To estimate the raise in serum iron, B12 and folate levels after 3 months of study salt consumption.

ELIGIBILITY:
Inclusion Criteria: • Willing to voluntarily participate in the study

* Can comprehend and comply with study requirements
* Aged between 18 and 45 years.
* No documented issues with child bearing potential
* Resident of the area of study for duration of study.
* Consume only study salt during study

Exclusion Criteria:

* Taking multivitamins or FA during study
* Pregnant or lactating at recruitment or during study
* Co-morbidities such as Malabsorption disorders, severe anemia (Hgb <8.0 g/dL), uncontrolled hypertension, (SBP ≥140 mm Hg or DBP ≥90 mm Hg), HIV, active TB or malaria infection
* History of prior SBA delivery
* Pre-existing medical conditions (i.e., cancer or need for regular medications)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of childbearing age who are non-lactating and willing to consume the study salt for the duration were recruited for voluntary participation into the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Measure changes in median serum folate levels between baseline and study endpoint | 2-6 months
  evaluate blood levels pre- and post-intake of study salt (fortified with folic acid)

CONTACTS AND LOCATIONS:
Overall Officials: Jogi Pattisapu, MD, Principal Investigator — Pediatric Neurosurgery
Locations (1):
- Pediatric Neurosurgery, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
redacted information will be made available upon request.

REFERENCES:
- [Derived] Pattisapu JV, Manda VV, Kottakki MNR, Kajana PM, Kancherla V, Bhaganagarapu HR, Veerappan V, Ediga A, Mannar V, Diosady L, Oakley GP Jr. Folic Acid-Fortified Iodized Salt and Serum Folate Levels in Reproductive-Aged Women of Rural India: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Mar 4;7(3):e241777. doi: 10.1001/jamanetworkopen.2024.1777. PMID 38457177